CLINICAL TRIAL: NCT00375219
Title: A Phase II Open-Label Study of the Subcutaneous Administration of Homoharringtonine. (Omacetaxine) (CGX-635) in the Treatment of Patients With Chronic Myeloid Leukemia. (CML) With the T315I BCR-ABL Gene Mutation
Brief Title: Homoharringtonine (Omacetaxine Mepesuccinate) in Treating Patients With Chronic Myeloid Leukemia (CML) With the T315I BCR-ABL Gene Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Collaborators: Cephalon (Industry); ChemGenex Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGX-635-CML-202; 2006-000176-32 (EudraCT Number)
Record Dates: First submitted 2006-09-08; First posted 2006-09-12 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Chronic Myeloid Leukemia; CML; HHT; Homoharringtonine; Omacetaxine; T315i; ChemGenex; ChemGenex Pharmaceuticals
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Homoharringtonine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- omacetaxine (Experimental): Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 3 years.
  Interventions: Drug: Omacetaxine mepesuccinate

INTERVENTIONS:
Drug: Omacetaxine mepesuccinate — Induction:
  1.25 mg/m^2 subcutaneously, twice daily for 14 consecutive days every 28 days until response. Patients not demonstrating evidence of clinical response after 6 induction cycles will be considered for removal from the study.
  Maintenance:
  1.25 mg/m^2 subcutaneously, twice daily for 7 consecutive days in a 28-day cycle, for up to 3 years.
  Other Names: Homoharringtonine; OMA; Synribo; HHT; CGX-635

SUMMARY:
To evaluate the safety and efficacy of subcutaneous administration of omacetaxine mepesuccinate (HHT) in achieving a clinical response in CML patients in chronic, accelerated, or blast phase who have failed prior imatinib therapy and have the T315I kinase domain gene mutation.

DETAILED DESCRIPTION:
Point mutations within the ABL kinase domain of the BCR-ABL gene are emerging as the most frequent mechanism for resistance to imatinib and resultant reactivation of kinase activity. The risk of mutation development is particularly high in patients who are beyond chronic phase, as well as those with a long duration of disease prior to imatinib therapy.

The T315I kinase domain (KD) point mutation has merited particular attention, as T315I expressing CML cells are markedly resistant to imatinib. CML patients with the T315I KD mutation, therefore, do not respond to continued treatment with imatinib, and preliminary clinical data indicate that neither of two newer tyrosine kinase inhibitors will have activity in patients with T315I KD mutation either.

Omacetaxine mepesuccinate (HHT) is a potent inducer of apoptosis (programmed cell death) in myeloid cells and inhibits angiogenesis (blood vessel formation). In Phase 2 studies, HHT has demonstrated clinical activity in patients with CML, both as a single agent and in-combination with other chemotherapeutic drugs. HHT works via a different mechanism than imatinib or other tyrosine kinase inhibitors (TKI's), and HHT has been shown to inhibit in vitro CML cell lines which harbor the T315I KD mutation and are highly resistant to imatinib. Therefore, CML patients who have the T315I KD mutation may still respond to treatment with HHT. HHT may therefore be an attractive therapeutic option for patients with the T315I KD mutation.

On this basis, a multicenter clinical trial is being conducted of HHT therapy for CML patients who have failed prior imatinib therapy and have the T315I KD mutation.

Patients will be treated with an induction course consisting of subcutaneous (SC) HHT twice daily for 14 consecutive days every 28 days. Patients who demonstrate a response, may receive maintenance therapy for up to 24 months, consisting of subcutaneous (SC) HHT twice daily for 7 days every 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, age 18 years or older
* Philadelphia chromosome (Ph) positive chronic myelogenous leukemia in either chronic, accelerated, or blast phase
* The patient will have the T315I BCR-ABL gene mutation
* Patients will have failed prior imatinib therapy
* ECOG performance status 0-2

Exclusion Criteria:

* NYHA class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia and requiring therapy, uncontrolled hypertension or congestive heart failure
* Myocardial infarction in the previous 12 weeks
* Lymphoid Ph+ blast crisis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-09-20 (Actual); Primary Completion 2010-03-23 (Actual); Study Completion 2013-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Cortes, MD, Principal Investigator — Univ. of Texas M.D. Anderson Cancer Center; Andreas Hochhaus, MD Prof Dr, Principal Investigator — Mannheim der Universitat Heidelberg
Locations (32):
- United States (10):
  - Teva Investigational Site 003, Los Angeles, California
  - Teva Investigational Site 007, Jacksonville, Florida
  - Teva Investigational Site 006, Atlanta, Georgia
  - Teva Investigational Site 008, Beech Grove, Indiana
  - Teva Investigational Site 011, Baltimore, Maryland
  - Teva Investigational Site 004, Boston, Massachusetts
  - Teva Investigational Site 005, Buffalo, New York
  - Teva Investigational Site 002, The Bronx, New York
  - Teva Investigational Site 010, Philadelphia, Pennsylvania
  - Teva Investigational Site 001, Houston, Texas
- Canada (2):
  - Teva Investigational Site 013, Montreal
  - Teva Investigational Site 009, Toronto
- France (10):
  - Teva Investigational Site 029, Bordeaux
  - Teva Investigational Site 021, Le Chesnay
  - Teva Investigational Site 022, Lille
  - Teva Investigational Site 020, Lyon
  - Teva Investigational Site 024, Nice
  - Teva Investigational Site 028, Paris
  - Teva Investigational Site 023, Poitiers
  - Teva Investigational Site 027, Strasbourg
  - Teva Investigational Site 025, Toulouse
  - Teva Investigational Site 026, Vandœuvre-lès-Nancy
- Germany (2):
  - Teva Investigational Site 031, Berlin
  - Teva Investigational Site 030, Mannheim
- Teva Investigational Site 050, Budapest, Hungary
- India (2):
  - Teva Investigational Site 071, Hyderabad
  - Teva Investigational Site 070, Mumbai
- Teva Investigational Site 090, Bologna, Italy
- Poland (2):
  - Teva Investigational Site 060, Gdansk
  - Teva Investigational Site 061, Warsaw
- Teva Investigational Site 080, Singapore, Singapore
- Teva Investigational Site 040, London, United Kingdom

REFERENCES:
- [Derived] Cortes J, Lipton JH, Rea D, Digumarti R, Chuah C, Nanda N, Benichou AC, Craig AR, Michallet M, Nicolini FE, Kantarjian H; Omacetaxine 202 Study Group. Phase 2 study of subcutaneous omacetaxine mepesuccinate after TKI failure in patients with chronic-phase CML with T315I mutation. Blood. 2012 Sep 27;120(13):2573-80. doi: 10.1182/blood-2012-03-415307. Epub 2012 Aug 15. PMID 22896000

RESULTS

PARTICIPANT FLOW:
Groups:
- CML: Chronic Phase: Study participants with chronic myeloid leukemia (CML) in the chronic phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 3 years.
- CML: Accelerated Phase: Study participants with chronic myeloid leukemia (CML) in the accelerated phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 3 years.
- CML: Blast Phase: Study participants with chronic myeloid leukemia (CML) in the blast phase at the time of enrollment. Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 3 years.
Period: Overall Study
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Started | 62 | 20 | 21
Completed | 3 | 0 | 0
Not Completed | 59 | 20 | 21
Not completed — Failure to achieve a response | 16 | 2 | 0
Not completed — Adverse Event | 8 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Request of Patient, PI, Sponsor or RA | 5 | 3 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Disease progression | 18 | 9 | 12
Not completed — Death | 4 | 3 | 7
Not completed — Hematologic resistance | 1 | 0 | 0
Not completed — Specific tyrosine kinase inhibitor avail | 1 | 0 | 0
Not completed — Allograft | 2 | 0 | 0
Not completed — Cord blood transplantation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent to treat population includes all participants who provide written informed consent and receive at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total
Number analyzed (Participants) | 62 | 20 | 21 | 103
Age, Continuous [Median (Full Range); unit: years] | 59 [26 to 83] | 59 [30 to 83] | 50 [19 to 64] | 57 [19 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 5 | 7 | 32
  Male | 42 | 15 | 14 | 71
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 48 | 12 | 13 | 73
  Black | 4 | 6 | 6 | 16
  Hispanic | 0 | 0 | 0 | 0
  Asian | 8 | 2 | 2 | 12
  Other | 2 | 0 | 0 | 2
Height [Median (Full Range); unit: centimeter] | 171.5 [146.0 to 192.0] | 172.0 [155.0 to 185.0] | 170.2 [157.0 to 196.0] | 171.0 [146.0 to 196.0]
Weight [Median (Full Range); unit: kilograms] | 77.7 [34.0 to 115.0] | 69.1 [40.0 to 118.8] | 68.8 [43.0 to 117.7] | 76.0 [34.0 to 118.8]
Body Surface Area (BSA) [Median (Full Range); unit: meters^2] | 1.9 [1.2 to 2.3] | 1.8 [1.3 to 2.3] | 1.8 [1.4 to 2.4] | 1.9 [1.2 to 2.4]
New York Heart Association (NYHA) Classification [Number; unit: participants] — * Class I: Cardiac disease, but no symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  * Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  * Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100 m). Comfortable only at rest.
  * Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bed-bound patients.
  participants
    Class I | 61 | 18 | 18 | 97
    Class II | 1 | 2 | 3 | 6
    Class III | 0 | 0 | 0 | 0
    Class IV | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group Performance Status [Number; unit: participants] — * Grade 0: Fully active, able to carry on all pre-disease activities without restriction;
  * Grade 1: Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  * Grade 2: Ambulatory and capable of all self-care but unable to work. Up and about more than 50% of waking hours;
  * Grade 3: Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  * Grade 4: Completely disabled. Cannot carry on any self-care. Confined to bed or chair.
  participants
    Grade 0 | 41 | 6 | 6 | 53
    Grade 1 | 20 | 11 | 9 | 40
    Grade 2 | 1 | 2 | 5 | 8
    Grade 3 | 0 | 1 | 1 | 2
Time from Initial Chronic Myeloid Leukemia (CML) Diagnosis [Median (Full Range); unit: months] | 50.0 [10.9 to 234.3] | 98.0 [34.3 to 285.6] | 46.6 [5.2 to 139.8] | 59.6 [5.2 to 285.6]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an Overall Hematologic Response by Subpopulation and Total Population
Description: Subpopulations reflect chronic myeloid leukemia (CML) phases at the time of enrollment: chronic, accelerated, and blast phase. Primary endpoints as adjudicated by the Data Monitoring Committee were used for the primary analyses.
  Overall hematologic response for chronic phase participants includes confirmed complete hematologic response (CHR). Overall hematologic response for accelerated or blast phase participants includes confirmed complete hematologic response (CHR), no evidence of leukemia (NEL), or return to chronic phase (RCP). Hematologic response must last >= 8 weeks to be considered meaningful.
  Response rates by disease phase were examined relative to an a priori value of 2.5% using a one-sided lower 95% exact binomial confidence limit. If the lower limit from the one-sided lower 95% confidence limit exceeds 2.5%, the observed response rate will have exceeded the minimum threshold required to demonstrate efficacy.
Time Frame: Day 1 up to 6 months
Population: Intent to treat population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total Participants: Treatment included induction therapy of subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 3 years.
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
percentage of participants | 77.4 [65.03 to NA] — Lower limit of the 2-sided 95% CI is reported | 55.0 [31.53 to NA] — Lower limit of the 2-sided 95% CI is reported | 9.5 [1.17 to NA] — Lower limit of the 2-sided 95% CI is reported | 59.2 [49.10 to NA] — Lower limit of the 2-sided 95% CI is reported

2. Primary Outcome: Percentage of Participants Achieving a Major Cytogenetic Response by Subpopulation and Total Population
Description: Subpopulations reflect chronic myeloid leukemia (CML) phases at the time of enrollment: chronic, accelerated, and blast phase. Primary endpoints as adjudicated by the Data Monitoring Committee were used for the primary analyses.
  Major cytogenetic response includes complete or partial response. Both confirmed and unconfirmed major cytogenetic response is considered meaningful.
  Unconfirmed response is based on a single bone marrow cytogenetic evaluation for participants where a confirmatory evaluation is not available.
  Complete response shows 0% Philadelphia chromosome positive (Ph+) cells. A partial response shows >0% - 35% Ph+ cells.
  Response rates by disease phase were examined relative to an a priori value of 2.5% using a one-sided lower 95% exact binomial confidence limit. If the lower limit from the one-sided lower 95% confidence limit exceeds 2.5%, the observed response rate will have exceeded the minimum threshold required to demonstrate efficacy.
Time Frame: Day 1 up to 6 months
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
percentage of participants | 22.6 [12.93 to NA] — Lower limit of the 2-sided 95% CI is reported | 5.0 [0.13 to NA] — Lower limit of the 2-sided 95% CI is reported | 0 [0 to 0] | 14.6 [8.39 to NA] — Lower limit of the 2-sided 95% CI is reported

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) by Subpopulation and Total
Description: TEAE are any untoward events that were newly occurring or worsening from Baseline.
  Treatment related toxicity was considered by the investigator to be unrelated, possibly, probably or unknown related to study drug.
  Severity was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v3.0 on the following scale: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death.
  A serious adverse event (SAE) is any untoward medical occurrence that is fatal or life-threatening; results in persistent or significant disability or incapacity; requires or prolongs in-patient hospitalization; is a congenital anomaly/birth defect in the offspring of a patient; and conditions not included in the above that may jeopardize the patient or may require intervention to prevent one of the outcomes listed above.
  A participant is only counted once in each category (at worst severity or strongest relationship).
Time Frame: up to 3 years
Population: Intent to treat
Measure: Number; unit: participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
participants
  >=1 TEAE | 61 | 20 | 21 | 102
  >= 1 SAE | 36 | 12 | 19 | 67
  Worst severity: Grade 1 | 0 | 1 | 0 | 1
  Worst severity: Grade 2 | 6 | 2 | 1 | 9
  Worst severity: Grade 3 | 9 | 4 | 4 | 17
  Worst severity: Grade 4 | 37 | 9 | 4 | 50
  Worst severity: Grade 5 | 9 | 4 | 12 | 25
  Relation to drug: Unrelated | 1 | 3 | 3 | 7
  Relation to drug: Possibly | 6 | 3 | 5 | 14
  Relation to drug: Probably | 54 | 13 | 13 | 80
  Relation to drug: Unknown | 0 | 1 | 0 | 1
  With hematologic toxicity | 55 | 13 | 13 | 81
  Discontinued treatment due to AE | 18 | 10 | 11 | 39
  Deaths during study or follow-up | 31 | 14 | 19 | 64
  Deaths during study (outcome of SAE) | 9 | 4 | 12 | 25

4. Secondary Outcome: Percentage of Participants in Each Cytogenetic Response Category Representing the Degree of Suppression of the Philadelphia Chromosome (Ph+)
Description: Cytogenetic response categories:
  * Complete: 0% Ph+ cells
  * Partial: >0%-35% Ph+ cells
  * Minor: >35%-65% Ph+ cells
  * Minimal: >65%-95% Ph+ cells
  * No Response: >95% Ph+ cells
  * Unevaluable: <20 metaphases were examined and/or response could not be assigned
Time Frame: Day 1 up to Month 9
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
percentage of participants
  Complete | 16.1 | 5.0 | 0 | 10.7
  Partial | 6.5 | 0 | 0 | 3.9
  Minor | 4.8 | 0 | 0 | 2.9
  Minimal | 16.1 | 5.0 | 9.5 | 12.6
  No Response | 37.1 | 30.0 | 38.1 | 35.9
  Unevaluable | 19.4 | 60.0 | 52.4 | 34.0

5. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) Representing the Degree of Suppression of BCR-ABL Transcript Levels Using the Housekeeping Gene GUS
Description: MMR is defined as a ratio of BCR-ABL/standard gene of less than 0.1% according to the international scale. BCR-ABL is a fusion gene of the breakpoint cluster region [BCR] gene and Abelson proto-oncogene [ABL] genes). This analysis used the standard gene GUS. Analysis was performed by quantitative reverse transcription polymerase chain reaction (qRT-PCR) of peripheral blood.
Time Frame: Day 1 up to Month 6
Population: Intent to treat population of participants who had evaluable samples. Participants with no data for these analyses either had degraded samples or the samples were missing.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 37 | 8 | 4 | 49
percentage of participants | 8.1 [1.7 to 21.9] | 12.5 [0.3 to 52.7] | 0 [NA to NA] — no participants met criteria | 8.2 [2.3 to 19.6]

6. Secondary Outcome: Percentage of Participants With Major Molecular Response (MMR) Representing the Degree of Suppression of BCR-ABL Transcript Levels Using the Housekeeping Gene ABL
Description: MMR is defined as a ratio of BCR-ABL/standard gene of less than 0.1% according to the international scale. BCR-ABL is a fusion gene of the breakpoint cluster region [BCR] gene and Abelson proto-oncogene [ABL] genes). This analysis used the standard gene ABL. Analysis was performed by quantitative reverse transcription polymerase chain reaction (qRT-PCR) of peripheral blood.
Time Frame: Day 1 up to Month 6
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 52 | 13 | 8 | 73
percentage of participants | 19.2 [9.6 to 32.5] | 15.4 [1.9 to 45.5] | 0 [NA to NA] — no participants met criteria | 16.4 [8.8 to 27.0]

7. Secondary Outcome: Percentage of Participants in Each Hematologic Response Category
Description: Complete Response (CHR)
  * Chronic phase must last at least 8 weeks: WBC <10*10^9/liter, platelets <450*10^9/liter, myelocytes + metamyelocytes <5% in blood, no blasts or promyelocytes in blood, <20% basophils in peripheral blood, no extramedullary involvement.
  * Accelerated and Blast phase must last at least 4 weeks: absolute neutrophil count 1.5*10^9/liter, platelets 100*10^9/liter, no blood blasts, bone marrow blasts <5%, no extramedullary disease.
  Partial Response - CHR plus one or more of the following:
  * Persistence of splenomegaly with a reduction of ≥50% from pre-treatment
  * Platelets > 450*10^9/L
  * Presence of immature cells in the peripheral blood
  * 5% to 25% blasts in the bone marrow
  * If extra-medullary disease pre-treatment, reduction by ≥50% Hematologic Improvement - CHR, except allowing persistent thrombocytopenia (<100*10^9/L), and a few immature cells No evidence of leukemia: Morphologic leukemia-free state, defined as <5% bone marrow blasts.
Time Frame: Day 1 up to Month 6
Population: Intent to treat
Measure: Number; unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
percentage of participants
  Complete response | 77.4 | 45.0 | 4.8 | 56.3
  Partial response | 0 | 0 | 0 | 0
  Hematologic improvement | 0 | 0 | 4.8 | 1.0
  Return to chronic phase | NA — Participants enrolled in chronic phase and therefore cannot respond (improve) to chronic phase. | 5.0 | 4.8 | 1.9
  No evidence of leukemia | NA — An overall hematologic response for chronic phase participants only included a complete hematologic response. | 5.0 | 0 | 1.0
  No response | 19.4 | 25.0 | 81.0 | 33.0
  Unevaluable | 3.2 | 20.0 | 4.8 | 6.8

8. Secondary Outcome: Percentage of Participants With Extramedullary Disease (EMD) at Baseline Achieving a Clinical Response
Description: Clinical response was defined by disease phase and based on evaluations by the independent Data Monitoring Committee (DMC).
  Chronic Phase subgroup: achieving a complete hematologic response and/or major cytogenetic response (complete cytogenetic response or partial cytogenetic response, confirmed or unconfirmed).
  Accelerated Phase and Blast Phase subgroups: achieving complete hematologic response, no evidence of leukemia, return to chronic phase, and/or major cytogenetic response (complete cytogenetic response or partial cytogenetic response, confirmed or unconfirmed).
  The percentage of participants achieving response with extramedullary disease at Baseline was to be summarized, if the sample size was sufficient. This analysis was not done as the sample was ultimately insufficient
Time Frame: Day 1 up to Month 9
Population: Intent to treat population of study participants who had extramedullary disease at baseline. Analysis not performed due to insufficient sample size.
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants With the Largest Percentage Reduction From Baseline of T315I Mutated BCR-ABL
Description: Summarization is based on the best of the individual response assessments. Not assessable indicates that the participant either had no baseline assessment or the % mutation could not be determined in the post-baseline assessment(s).
Time Frame: Day 1 up to Month 9
Population: Intent to treat population of participants with post-baseline assessment of T315I mutated BCR ABL
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 50 | 13 | 8 | 71
percentage of participants
  100% reduction | 6.0 [2.0 to 25.0] | 0 [0 to 0] | 0 [0 to 0] | 4.2 [1.3 to 17.5]
  75-99% reduction | 4.0 [0.8 to 20.8] | 0 [0 to 0] | 25.0 [4.3 to 77.7] | 5.6 [2.4 to 20.4]
  50-74% reduction | 14.0 [9.3 to 40.0] | 0 [0 to 0] | 12.5 [0.4 to 64.1] | 11.3 [7.7 to 30.8]
  25-49% reduction | 18.0 [13.8 to 46.8] | 15.4 [2.8 to 60.0] | 0 [0 to 0] | 15.5 [12.3 to 38.0]
  1-24% reduction | 8.0 [3.5 to 29.0] | 38.5 [21.2 to 86.3] | 12.5 [0.4 to 64.1] | 14.1 [10.7 to 35.7]
  0% reduction | 14.0 [9.3 to 40.0] | 15.4 [2.8 to 60.0] | 25.0 [4.3 to 77.7] | 15.5 [12.3 to 38.0]
  Not assessable | 36.0 [NA to NA] — 95% CI not calculated for a non-response category. | 30.8 [NA to NA] — 95% CI not calculated for a non-response category. | 25.0 [NA to NA] — 95% CI not calculated for a non-response category. | 33.8 [NA to NA] — 95% CI not calculated for a non-response category.

10. Secondary Outcome: Number of Treatment Cycles Needed to Achieve Best Hematologic Response
Description: Induction therapy was administered for 14 consecutive days for each 28 days cycle, for up to 6 cycles. All treatment arms were given omacetaxine mepesuccinate via subcutaneous (SC) administration at 1.25 mg/m^2 twice a day (BID) for the 14 consecutive days.
Time Frame: Day 1 up to Month 6
Population: Intent to treat population of participants who had a response to treatment
Measure: Median (Full Range); unit: treatment cycles
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 48 | 11 | 2 | 61
treatment cycles | 1.0 [1 to 5] | 1.0 [1 to 3] | 1.0 [1 to 1] | 1.0 [1 to 5]

11. Secondary Outcome: Number of Treatment Cycles Needed to Achieve Best Cytogenetic Response
Time Frame: Day 1 up to 22 months
Population: Intent to treat population of participants who had a cytogenetic response
Measure: Median (Full Range); unit: treatment cycles
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 27 | 2 | 2 | 31
treatment cycles | 3.0 [1 to 22] | 2.5 [2 to 3] | 2.0 [1 to 3] | 3.0 [1 to 22]

12. Secondary Outcome: Kaplan-Meier Estimates for Time to Onset of Best Hematologic Response
Description: Time to onset was analyzed using Kaplan-Meier estimates. Participants who did not achieve a response are censored at their last visit day.
  Overall hematologic response for chronic phase participants includes confirmed complete hematologic response (CHR). Overall hematologic response for accelerated or blast phase participants includes confirmed complete hematologic response (CHR), no evidence of leukemia (NEL), or return to chronic phase (RCP). Hematologic response must last >= 8 weeks to be considered meaningful.
Time Frame: Day 1 up to Month 6
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 62 | 20 | 21
months | 0.46 [0.39 to 0.92] | 1.74 [0.00 to NA] — A large percentage of participants were censored. | NA [NA to NA] — A large percentage of participants were censored.

13. Secondary Outcome: Kaplan-Meier Estimates for Time to Onset of Best Cytogenetic Response
Description: Time to onset was analyzed using Kaplan-Meier estimates. Participants who did not achieve a response are censored at their last visit day.
  Major cytogenetic response includes complete or partial response. Both confirmed and unconfirmed major cytogenetic response is considered meaningful.
  Unconfirmed response is based on a single bone marrow cytogenetic evaluation for participants where a confirmatory evaluation is not available.
  Complete response shows 0% Philadelphia chromosome positive (Ph+) cells. A partial response shows >0% - 35% Ph+ cells.
Time Frame: up to 3 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 62 | 20 | 21
months | NA [NA to NA] — A large percentage of participants were censored. | NA [NA to NA] — A large percentage of participants were censored. | NA [NA to NA] — A large percentage of participants were censored.

14. Secondary Outcome: Kaplan-Meier Estimates for Duration of Best Hematologic Response
Description: Duration of response is defined as the time from first reported date of hematologic response until the earliest date of objective evidence of disease progression, relapse or death. Data was censored at the last examination date for participants with ongoing response or participants who discontinued treatment for reasons other than adverse event, disease progression or death.
Time Frame: up to 4 years
Population: Intent to treat population of participants who had a response
Measure: Median (Full Range); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 48 | 11 | 2
months | 9.08 [1.61 to 71.38] | 3.59 [1.25 to 25.46] | 3.31 [1.68 to 4.93]

15. Secondary Outcome: Kaplan-Meier Estimates for Duration of Best Cytogenetic Response
Description: Duration of response is defined as the time from first reported date of cytogenetic response until the earliest date of objective evidence of disease progression, relapse or death. Data was censored at the last examination date for participants with ongoing response or participants who discontinued treatment for reasons other than adverse event, disease progression or death.
Time Frame: up to 4 years
Population: Intent to treat population of participants who had a response
Measure: Median (Full Range); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase
Number analyzed (Participants) | 14 | 1 | 0
months | 6.64 [2.34 to 59.38] | 16.35 [16.35 to 16.35] |

16. Secondary Outcome: Kaplan-Meier Estimates for Time to Disease Progression
Description: Time to disease progression is defined as the time from the initiation of treatment until the onset date of death, the development of CML accelerated phase or blast phase, or the loss of complete hematologic response or major cytogenetic response, whichever came first. Participants were censored only if they did not have progression or if they discontinued treatment for reasons other than AE, progression or death.
Time Frame: up to 4 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
months | 7.73 [5.79 to 11.02] | 4.74 [1.81 to 9.01] | 2.20 [1.48 to 3.26] | 5.86 [3.88 to 7.04]

17. Secondary Outcome: Kaplan-Meier Estimates for Overall Survival
Description: Overall survival is defined as the time from the initiation of treatment until death from any cause or the last day of participant contact or evaluation for participants that were lost to follow-up. Participants were censored t the last recorded contract or evaluation when a participant was alive at time of analysis. A quarterly phone survey was conducted to collect survival data for participants who discontinued from the study.
Time Frame: up to 4 years
Population: Intent to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CML: Chronic Phase | CML: Accelerated Phase | CML: Blast Phase | Total Participants
Number analyzed (Participants) | 62 | 20 | 21 | 103
months | 49.31 [24.97 to NA] — A large percentage of participants were censored | 18.72 [4.74 to 32.07] | 3.45 [2.20 to 4.84] | 21.51 [12.01 to 36.88]

ADVERSE EVENTS:
Time Frame: up to 4 years
Groups:
- Omacetaxine: Treatment was the same for all cohorts: induction therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 14 consecutive days every 28 (±3) days for up to 6 cycles. Maintenance therapy was subcutaneous (SC) administration of omacetaxine at 1.25 mg/m^2 twice a day (BID), administered for 7 consecutive days every 28 (±3) days for up to 24 months.
Arm/Group | Omacetaxine
Serious Adverse Events (participants affected / at risk) | 67/103
Other Adverse Events (participants affected / at risk) | 100/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine (N=103)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Bone marrow failure (Blood and lymphatic system disorders) | 8 (10)
Bone marrow necrosis (Blood and lymphatic system disorders) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 12 (14)
Haematotoxicity (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1)
Leukostasis (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (4)
Pancytopenia (Blood and lymphatic system disorders) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (17)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Chromosomal deletion (Congenital, familial and genetic disorders) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Aplasia (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Disease progression (General disorders) | 12 (12)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 3 (3)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Leukaemic infiltration extramedullary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 2 (2)
Convulsion (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Renal failure chronic (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omacetaxine (N=103)
Anaemia (Blood and lymphatic system disorders) | 56 (196)
Bone marrow failure (Blood and lymphatic system disorders) | 8 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 15 (21)
Leukocytosis (Blood and lymphatic system disorders) | 10 (20)
Leukopenia (Blood and lymphatic system disorders) | 18 (64)
Lymphopenia (Blood and lymphatic system disorders) | 13 (39)
Neutropenia (Blood and lymphatic system disorders) | 48 (139)
Pancytopenia (Blood and lymphatic system disorders) | 15 (22)
Thrombocytopenia (Blood and lymphatic system disorders) | 67 (253)
Tachycardia (Cardiac disorders) | 8 (8)
Abdominal pain (Gastrointestinal disorders) | 14 (26)
Abdominal pain upper (Gastrointestinal disorders) | 14 (16)
Constipation (Gastrointestinal disorders) | 18 (18)
Diarrhoea (Gastrointestinal disorders) | 40 (107)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Gingival bleeding (Gastrointestinal disorders) | 8 (9)
Mouth ulceration (Gastrointestinal disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 36 (96)
Vomiting (Gastrointestinal disorders) | 15 (17)
Asthenia (General disorders) | 22 (59)
Chest pain (General disorders) | 7 (10)
Chills (General disorders) | 7 (7)
Disease progression (General disorders) | 18 (19)
Fatigue (General disorders) | 35 (65)
Injection site bruising (General disorders) | 8 (8)
Injection site erythema (General disorders) | 17 (66)
Injection site pain (General disorders) | 8 (10)
Injection site reaction (General disorders) | 7 (7)
Mucosal inflammation (General disorders) | 6 (8)
Oedema peripheral (General disorders) | 20 (30)
Pyrexia (General disorders) | 30 (36)
Hyperbilirubinaemia (Hepatobiliary disorders) | 7 (17)
Oral herpes (Infections and infestations) | 7 (8)
Pneumonia (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 11 (15)
Contusion (Injury, poisoning and procedural complications) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 12 (12)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 10 (20)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (39)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 12 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (19)
Dizziness (Nervous system disorders) | 8 (9)
Headache (Nervous system disorders) | 15 (26)
Anxiety (Psychiatric disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 14 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (15)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (25)
Alopecia (Skin and subcutaneous tissue disorders) | 14 (14)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (10)
Erythema (Skin and subcutaneous tissue disorders) | 6 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 6 (9)
Petechiae (Skin and subcutaneous tissue disorders) | 7 (8)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (10)
Rash (Skin and subcutaneous tissue disorders) | 15 (20)
Haematoma (Vascular disorders) | 7 (7)
Hypertension (Vascular disorders) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.